CLINICAL TRIAL: NCT02989740
Title: Combined Optical Coherence Tomography Morphologic and Fractional Flow Reserve Hemodynamic Assessment of Non-Culprit Lesions to Better Predict Adverse Event Outcomes in Diabetes Mellitus Patients. COMBINE (OCT-FFR) Prospective Register
Brief Title: Optical Coherence Tomography Morphologic and Fractional Flow Reserve Assessment in Diabetes Mellitus Patients
Acronym: COMBINE
Status: Completed | Type: Observational
Sponsor: Diagram B.V. (Other)
Collaborators: Isala (Other); St. Jude Medical Nederland B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: 9241
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease; Coronary Atheroscleroses
Keywords: Diabetes Mellitus; Thincap fibroatheroma; Optical Coherence Tomography; Fractional Flow Reserve
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Patients with negative FFR (> 0.80) in the target lesion & decided on OCT (Optical Coherence Tomography) imaging findings with NO thin-cap fibroatheroma
  Interventions: Procedure: Optical Coherence Tomography
- Group B: Patients with negative FFR (> 0.80) in the target lesion & decided on OCT (Optical Coherence Tomography) imaging findings presence of ≥ thin-cap fibroatheroma
  Interventions: Procedure: Optical Coherence Tomography
- Group C: Patients hosting FFR-positive target lesions that have been treated with PCI as per standard care and have further no TCFA lesions.
  Interventions: Procedure: Optical Coherence Tomography

INTERVENTIONS:
Procedure: Optical Coherence Tomography — Patients aged ≥ 18 years bearing target lesions that fulfil the inclusion criteria and have undergone FFR and OCT imaging as per clinical practice will be enrolled in the study.
  Other Names: OCT

SUMMARY:
Title:

Combined Optical Coherence Tomography Morphologic and Fractional Flow Reserve Hemodynamic Assessment of Non-Culprit Lesions to Better Predict Adverse Event Outcomes in Diabetes Mellitus Patients COMBINE (OCT-FFR) Prospective Register

To study the natural evolution of patients with at least one intermediate angiographic but non-hemodynamic significant stenotic lesion, in two subgroups of patients, with TCFA vs. no TCFA as detected by OCT imaging and to compare these two groups of patients with each other as well as to a subset of patients with FFR-positive and PCI-treated intermediate lesions on future MACE.

DETAILED DESCRIPTION:
Hypothesis Diabetes Mellitus (DM) patients with angiographically intermediate coronary lesions remain at risk for future MACE events, including those patients with fractional flow reserve (FFR) negative lesions. Use of FFR measurements combined with Optimal Coherence Tomography (OCT) detection of thin-cap fibroatheroma (TCFA) in will help predict future MACE rates.

Objective To study the natural evolution of patients with at least one intermediate angiographic but non-hemodynamic significant stenotic lesion, in two subgroups of patients, with TCFA vs. no TCFA as detected by OCT imaging and to compare these two groups of patients with each other as well as to a subset of patients with FFR-positive and PCI-treated intermediate lesions on future MACE.

Design Prospective, open label natural history registry. DM patients bearing target lesions {Any de novo lesion with an angiographic visual estimation of ≥ 40%- ≤ 80% Diameter Stenosis (DS) that is located in a non-grafted coronary segment. In patients with an MI at presentation the target lesion should be different from the culprit lesion} and have undergone FFR and OCT imaging as for clinical routine will be prospectively enrolled and followed. Patients with negative FFR (> 0.80) will be divided in two categories depending on corelab OCT imaging findings: No-TCFA (cap thickness >65µ) (Group A) or TCFA (cap thickness ≤ 65µ) (group B). All patients that had a positive FFR and therefore have been treated with PCI as per standard care in all target lesions will also be followed (group C), however if after the PCI there is at least one remaining target lesion where FFR was negative these patients should be followed in group A or B depending on the OCT findings. Clinical endpoints at 1.5 year will be recorded.

The investigators strongly recommend that all major epicardial coronary vessels of stentable size that show any form of atherosclerosis to be interrogated with FFR and OCT.

The investigators strongly recommend to not perform cap thickness measurements in the cathlab. The plaque cap thickness as measured in the corelab will not be disclosed to operators and patients.

Population Patients aged ≥18 years Diabetes mellitus (DM) patients with any presentation. Coronary angiography, FFR and OCT imaging in at least one coronary de novo stenosis in a native vessel with a visually estimated diameter of stenosis (DS) of ≥ 40%-≤ 80% (target lesion).

Angiographic criteria target lesion:

(i) ≥ 40%-≤ 80% diameter stenosis (DS) (ii) de novo lesion located in native non-grafted vessel (iii) target lesion reference diameter of ≥ 2.0 mm (iv) TIMI 3 flow

Primary Endpoint The per patient incidence of the target lesion(s) related composite MACE defined as Cardiac Death, MI, clinically-driven target lesion revascularisation or hospitalization due to unstable or progressive angina at 18 months in the FFR-negative No-TCFA (Group A) and FFR-negative TCFA (Group B).

Statistics This is an observational study (prospective natural history register) where no randomization takes place, therefore a power calculation is strictly not necessary.

However, in order to observe meaningful differences between groups (as described in the design) and deduct founded conclusions, the minimal number of patients required was calculated as follows. The target lesion related primary endpoint at 18 months in the A and B group respectively are assumed to be 5 % and 20% respectively. Taking into account an expected loss in FU of 7%, a total of 500 patients enrolled in the study will provide 80% power to reject the null hypothesis with 5% type I error (alpha). The enrolment in group C will stop after the first 166 patients have been enrolled in this group. The rest of the rest of 334 patients will be distributed in groups A and B depending on the OCT corelab findings. Nul hypothesis: the MACE rate in group B is not different from group A.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. History of DM with any indication for angiography (Stable Angina (SA) or any type of Acute Coronary Syndrome (ACS) including ST-Elevation MI).
3. Coronary angiography, including FFR and OCT imaging of at least one coronary de novo stenosis in a native not-grafted vessel with a visually estimated diameter stenosis (DS) of ≥ 40 - ≤ 80% (target lesion) . Target lesion should be other than the culprit lesion(s) in patients presenting with MI (STEMI or non-STEMI).

Exclusion Criteria:

1. TIMI flow < 3 in the target lesion(s)
2. Target lesion reference diameter (on visual estimation) < 2.0 mm
3. Known left ventricular ejection fraction <30%
4. Known malignancy
5. Life expectancy < 2 years
6. Unwilling or unable to provide inform consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The COMBINE (OCT-FFR) Trial is an investigator driven study: a prospective natural history registry. Patients aged ≥ 18 years bearing target lesions (see definition section) that fulfil the inclusion criteria and have undergone FFR and OCT imaging as per clinical practice will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
The per patient incidence of the target lesion(s) related composite MACE | 18 months after procedure
  The per patient incidence of the target lesion(s) related composite MACE defined as Cardiac Death, MI, clinically-driven target lesion revascularisation or hospitalization due to unstable or progressive angina at 18 months in the FFR-negative No-TCFA (Group A) and FFR-negative TCFA (Group B).

SECONDARY OUTCOMES:
The per patient incidence of the target lesion(s) related composite MACE: | 18 months after procedure
  Cardicac death, MI, clinically- driven revascularization or hospitalization due to unstable or progressive angina between FFR-negative TCFA (Group B) and the group of patients with PCI-treated FFR-positive lesions (Group C).
The per patient incidence composite MACE | 18 months after procedure
  The per patient incidence composite MACE: Cardiac death, MI, any clinically driven-revascularization or hospitalization due to unstable or progressive angina between FFR-negative TCFA (Group B) and the group of patients with PCI treated FFR positive lesions (Group C).
The incidence of MACE (Cardiac death, MI, any clinically driven-revascularization or hospitalization due to unstable or progressive angina) | 18 months after procedure
  deriving from non PCI treated lesions between TCFA hosting patients anywhere in the major coronary of stentable size vs. patients with no TCFA (this analysis will be run in the total pool of patients after treatment of all FFR positive lesions and does not take in account the angiographic severity of the lesions ie. the location of the TCFA can be elsewhere than the target lesion )

CONTACTS AND LOCATIONS:
Overall Officials: E Kedhi, MD PhD, Principal Investigator — Erasmus Academical Hospital Brussels
Locations (1):
- Isala, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kennedy MW, Fabris E, Ijsselmuiden AJ, Nef H, Reith S, Escaned J, Alfonso F, van Royen N, Wojakowski W, Witkowski A, Indolfi C, Ottervanger JP, Suryapranata H, Kedhi E. Combined optical coherence tomography morphologic and fractional flow reserve hemodynamic assessment of non- culprit lesions to better predict adverse event outcomes in diabetes mellitus patients: COMBINE (OCT-FFR) prospective study. Rationale and design. Cardiovasc Diabetol. 2016 Oct 10;15(1):144. doi: 10.1186/s12933-016-0464-8. PMID 27724869
- [Result] Kedhi E, Berta B, Roleder T, Hermanides RS, Fabris E, IJsselmuiden AJJ, Kauer F, Alfonso F, von Birgelen C, Escaned J, Camaro C, Kennedy MW, Pereira B, Magro M, Nef H, Reith S, Al Nooryani A, Rivero F, Malinowski K, De Luca G, Garcia Garcia H, Granada JF, Wojakowski W. Thin-cap fibroatheroma predicts clinical events in diabetic patients with normal fractional flow reserve: the COMBINE OCT-FFR trial. Eur Heart J. 2021 Dec 1;42(45):4671-4679. doi: 10.1093/eurheartj/ehab433. PMID 34345911
- [Derived] Wang Z, Kedhi E, Liu X, Li C, Huang J, Zhong J, Qu X, Wijns W, Tu S; COMBINE OCT-FFR Study Group. Prognostic Implications of Angiographically Derived Coronary Radial Wall Strain in Diabetic Patients and Non-Flow-Limiting Stenosis. JACC Cardiovasc Interv. 2025 May 26;18(10):1232-1242. doi: 10.1016/j.jcin.2025.02.009. Epub 2025 May 10. PMID 40347200
- [Derived] Volleberg RHJA, Rroku A, Mol JQ, Hermanides RS, van Leeuwen M, Berta B, Meuwissen M, Alfonso F, Wojakowski W, Belkacemi A, Roleder T, Kedhi E, van Royen N; COMBINE (OCT-FFR) and PECTUS-obs investigators. FFR-Negative Nonculprit High-Risk Plaques and Clinical Outcomes in High-Risk Populations: An Individual Patient-Data Pooled Analysis From COMBINE (OCT-FFR) and PECTUS-obs. Circ Cardiovasc Interv. 2025 Feb;18(2):e014667. doi: 10.1161/CIRCINTERVENTIONS.124.014667. Epub 2025 Jan 22. PMID 39840429
- [Derived] Del Val D, Berta B, Roleder T, Malinowski K, Bastante T, Hermanides RS, Wojakowski W, Fabris E, Cuesta J, De Luca G, Rivero F, Alfonso F, Kedhi E. Vulnerable plaque features and adverse events in patients with diabetes mellitus: a post hoc analysis of the COMBINE OCT-FFR trial. EuroIntervention. 2024 Jun 3;20(11):e707-e717. doi: 10.4244/EIJ-D-23-00628. PMID 38840580
- [Derived] Fabris E, Berta B, Hommels T, Roleder T, Hermanides RS, Rivero F, von Birgelen C, Escaned J, Camaro C, Kennedy MW, Pereira B, Magro M, Nef H, Reith S, Roleder-Dylewska M, Gasior P, Malinowski KP, De Luca G, Garcia-Garcia HM, Granada JF, Wojakowski W, Kedhi E. Long-term outcomes of patients with normal fractional flow reserve and thin-cap fibroatheroma. EuroIntervention. 2023 Feb 6;18(13):e1099-e1107. doi: 10.4244/EIJ-D-22-00306. PMID 36170036
- [Derived] Fabris E, Berta B, Roleder T, Hermanides RS, IJsselmuiden AJJ, Kauer F, Alfonso F, von Birgelen C, Escaned J, Camaro C, Kennedy MW, Pereira B, Magro M, Nef H, Reith S, Roleder-Dylewska M, Gasior P, Malinowski K, De Luca G, Garcia-Garcia HM, Granada JF, Wojakowski W, Kedhi E. Thin-Cap Fibroatheroma Rather Than Any Lipid Plaques Increases the Risk of Cardiovascular Events in Diabetic Patients: Insights From the COMBINE OCT-FFR Trial. Circ Cardiovasc Interv. 2022 May;15(5):e011728. doi: 10.1161/CIRCINTERVENTIONS.121.011728. Epub 2022 Apr 29. PMID 35485232
- See also: Cardiovascular Diabetology — http://cardiab.biomedcentral.com/articles/10.1186/s12933-016-0464-8